CLINICAL TRIAL: NCT04864678
Title: Vaccination Coverage and Uptake in Young People Experiencing or at Risk of Homelessness
Status: Completed | Type: Observational
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: RCH League of Former Trainees and Associates Inc (Unknown); Royal Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 60835
Record Dates: First submitted 2021-01-28; First posted 2021-04-29 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Homeless Youth
Keywords: homeless youth; vaccination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young people who are experiencing or at risk of homelessness: Young people aged 15-24 years who have accessed a homeless youth service, refuge, or flexible learning center in Melbourne, Australia.
  Interventions: Other: Referral to the Young People's Health Service immunisation nurse

INTERVENTIONS:
Other: Referral to the Young People's Health Service immunisation nurse — Young people who have been referred to an immunisation nurse at the Young People's Health Service.

SUMMARY:
This retrospective audit will investigate if young people who are homeless or at risk of homelessness in Melbourne were up-to-date with routine childhood and adolescent vaccines on first encounter with a nurse-led primary health clinic (the Young People's Health Service), and if they commenced and completed immunisation catch-up plans following referral to the Young People's Health Service immunisation nurse.

The purpose of the proposed study is to establish baseline immunisation coverage within the targeted population, then to explore the impact of an immunisation nurse role on immunisation coverage in a population of young people aged 15-24 years who are experiencing or at risk of homelessness.

The Young People's Health Service is a program of the Royal Children's Hospital Department of Adolescent Medicine. The data collected will be sourced solely from the Royal Children's Hospital Electronic Medical Records.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 15-24 years inclusive at enrolment
* Has a signed general consent/referral form to the Young People's Health Service immunisation nurse between 19th February 2019 - 19th July 2020 and scanned into their EMR. Verbal consent is accepted.
* Was referred from a clinic or outreach location attended by the Young People's Health Service (i.e. a service for people experiencing homelessness)

Exclusion Criteria:

* Does not have a signed consent/referral form to Young People's Health Service immunisation nurse

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young people aged 15-24 years of all genders who have been referred to the Young People's Health Service immunisation nurse will be included. They have accessed a homeless youth service, refuge, or flexible learning centre in Melbourne, Australia. The study will include those who were referred between 19th February 2019 to 19th July 2020.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants referred to the Young People's Health Service immunisation nurse who were up-to-date for their age for vaccines on both the National Immunisation Program and the Victorian State Government Schedule. | Participants who were referred to the Young People's Health Service between the study time period (Between 19th February 2019 - 19th May 2021)
  Young people who meet eligibility criteria will be considered up-to-date on referral if their immunisation history statement at the time of referral meets the criteria to be considered up to date as detailed in Appendix II in the Study Protocol.
  The percentage of the young people in the population who are up-to-date for their age with each vaccine will be described.
Proportion of participants referred to the Young People's Health Service immunisation nurse who were are at increased risk of vaccine-preventable diseases. | All available medical records for the participant on the Royal Children's Hospital Electronic Medical Records regardless of time frame
  Where available, data collected from the Electronic Medical Records (EMR) will include risk factors for vaccine-preventable diseases and relevant social determinants of health based on the Australian Institute of Health and Welfare, the Australian Government Department of Health and the National Centre for Immunisation Research and Surveillance publications.
  Participants will be considered at increased risk of vaccine-preventable diseases if the EMR includes documentation of at least one of: a history of identifying as Aboriginal or Torres Strait Islander, of arriving in Australia as a migrant, refugee or asylum seeker, of incarceration, of men who have sex with men, of alcohol or other drug misuse, of smoking cigarettes, of living with Hepatitis C or HIV, of out of home care, of being a young parent, of having non-professional tattoos, or of sex work.

SECONDARY OUTCOMES:
Proportion of participants referred to the Young People's Health Service immunisation nurse who commence a vaccine catch-up plan. | Between 19th February 2019 - 19th May 2021
  Electronic medical records will be reviewed to record the percentage of participants who were not up-to-date with scheduled vaccines for their age on referral, and commenced a vaccine catch-up plan following referral to an immunisation nurse at the Young People's Health Service.
  Vaccines required to complete a vaccine catch-up plan will depend on the age of the participant and will be determined by an immunisation nurse.
  A participant will be considered to have commenced an immunisation catch-up plan if they receive at least one immunisation on the plan.
Proportion of participants referred to the Young People's Health Service immunisation nurse who complete a vaccine catch-up plan. | Between 19th February 2019 - 19th May 2021
  Electronic medical records will be reviewed to record the percentage of participants who were not up-to-date with scheduled vaccines for their age, and completed a vaccine catch-up plan following an encounter with an immunisation nurse at the Young People's Health Service.
  Vaccines required to complete a vaccine catch-up plan will depend on the age of the participant and will be determined by an immunisation nurse.
  A participant will be considered to have completed an immunisation catch-up plan if they receive all immunisations on the plan.
Mean number of follow-up contact attempts (all types) sent to young people attending the Young People's Health Service per immunisation visit. | Between 19th February 2019 - 19th May 2021
  The mean number of contact attempts sent by staff of the Young People's Health Service to young people who require immunisation catch-up visits. Contact attempts include SMS, email, phone call, in person reminder, and letter.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda L Tominc, MNSc, Principal Investigator — Royal Children's Hospital
Locations (1):
- The Royal Children's Hospital Melbourne, Parkville, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided